CLINICAL TRIAL: NCT01288222
Title: KIR Genotyping for Unrelated Donor (URD) Selection Prior to Hematopoietic Cell Transplantation (HCT) for AML: Selecting a Favorable KIR Donor
Brief Title: Selecting a Favorable KIR Donor in Unrelated HCT for AML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010LSUC043; MT2010-06 (Other: Blood and Marrow Transplantation Program); P01CA111412 (NIH)
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: acute myelogenous leukemia; hematopoietic cell transplantation; unrelated donor
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unrelated Donor Transplant Patients (Experimental): Patients with acute myeloid leukemia who have received KIR genotype from an unrelated donor transplant.
  Interventions: Other: KIR genotype

INTERVENTIONS:
Other: KIR genotype — KIR genotype data from unrelated donor are collected

SUMMARY:
Donors with favorable KIR B haplotype gene content have yielded reduced relapse risk and improved leukemia free survival (LFS) in retrospective analyses of unrelated donor (URD) hematopoietic cell transplantation (HCT) for acute myelogenous leukemia (AML). Specifically, donors with more KIR B gene content and those who are homozygous for the centromeric (Cen) B haplotype genes (as opposed to the telomeric (Tel) genes confer the most protective effect. This study proposes to prospectively test and validate the utility and effectiveness of further informing URD identification and selection by KIR genotyping as a supplement to HLA matching and the other variables known or suspected to indicate the best URD for a patient.

Hypotheses:

1. Favorable KIR donors will improve protection against relapse and improve leukemia free survival (LFS) after URD HCT for AML.
2. Directed study procedures for rapid KIR genotyping and reporting to searching Transplant Centers (TC) can inform donor search and selection without delay in donor availability for HCT.

DETAILED DESCRIPTION:
Transplant Centers will select the best HLA matched, and as appropriate, preferred KIR donor.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute myeloid leukemia (AML) undergoing screening for potential URD HCT
* Potential URD undergoing screening to provide a HCT graft to a patient with acute myeloid leukemia (AML) at a participating institution
* Provides written consent

Exclusion Criteria:

Transplant Centers will select the best HLA matched, and as appropriate, preferred KIR donor. In situations where the preferred (best > better > neutral) KIR donor is not selected in favor of a less favorable KIR genotype donor, the center will report one or more defined reasons (donor age; gender; parity; CMV status; ABO status; availability/logistics; other) for the choice (among equivalently HLA matched donors).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Relapse | 2 Years
  To measure the impact of donor selection for KIR genotype in allogeneic URD HCT for AML on cumulative incidence of relapse. We will determine a quantitative estimate of the likelihood of better KIR donors identified with routine, non-directed donor selection along with KIR genotyping data. The observed incidence of success in a better KIR donor identified within 8 weeks will be compared to the original donor genotype expected frequencies identified in our retrospective genotyping of 1086 donors selected for AML transplants.

SECONDARY OUTCOMES:
Incidence of Relapse-Free Survival | 2 Years
Overall Survival | 2 Years
Incidence of Engraftment | 2 Years
Incidence of Graft Versus Host Disease | 2 Years
Incidence of Transplant Related Mortality | 2 Years
  Number of patients who died within 2 years of transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weisdorf, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (19):
- United States (19):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center Cancer Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Kansas University Cancer Center, Kansas City, Kansas
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Presbyterian Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Sammons Cancer Center, Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Cooley S, Weisdorf DJ, Guethlein LA, Klein JP, Wang T, Marsh SG, Spellman S, Haagenson MD, Saeturn K, Ladner M, Trachtenberg E, Parham P, Miller JS. Donor killer cell Ig-like receptor B haplotypes, recipient HLA-C1, and HLA-C mismatch enhance the clinical benefit of unrelated transplantation for acute myelogenous leukemia. J Immunol. 2014 May 15;192(10):4592-600. doi: 10.4049/jimmunol.1302517. Epub 2014 Apr 18. PMID 24748496